CLINICAL TRIAL: NCT02706236
Title: A Single-Center Prospective Randomized Placebo Controlled Trial of Pancreatic Enzyme Supplements (Pancrelipase) for Treating Pain in Patients With Chronic Pancreatitis
Brief Title: Trial of Pancreatic Enzyme Supplements (Pancrelipase) for Treating Pain in Patients With Chronic Pancreatitis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no funding was awarded
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Timothy Gardner, Associate Professor of Medicine, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: D16084
Record Dates: First submitted 2016-02-27; First posted 2016-03-11 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Pancrelipase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Arm (Active Comparator): Pancreatic enzyme replacement (Pancrelipase) with meals and snacks daily, for 4 weeks.
  Interventions: Drug: Pancrelipase
- Placebo Arm (Placebo Comparator): Lactose placebo tablets with meals and snacks, for 4 weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Pancrelipase — Oral Pancrelipase, 720,000 units spread throughout the day with meals and snacks, taken daily PO for 4 weeks
  Arms: Intervention Arm
Drug: placebo — Placebo will consist of lactose, spread throughout the day with meals and snacks, taken daily PO for 4 weeks
  Arms: Placebo Arm

SUMMARY:
The study purpose is to characterize the effect of pancreatic enzyme supplementation on chronic pancreatitis type pain.

DETAILED DESCRIPTION:
Study Type: Interventional, randomized, double-blind, placebo-controlled, crossover design, efficacy study Intervention arm: Pancreatic enzyme replacement (Pancrelipase) with meals and snacks daily, for 4 weeks.

Placebo arm: Lactose placebo tablets with meals and snacks, for 4 weeks. Washout Phase: Weeks 4 to 6, there will be cessation of placebo or Pancrelipase use.

Crossover Phase: Weeks 6 to 10, initial placebo arm receives Pancrelipase, Pancrelipase arm receives placebo

Surveys - Izbicki score and PANQOLI assessment occur at Week 0, 4, 6, and 10. Narcotic and non-narcotic usage will also be noted at these intervals. Patient will also report the tobacco and alcohol use.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic pancreatitis based on chronic pancreatitis-type pain > 6 months leading to impaired quality of life AND at least 1 of the following (27):
* Confirmed diagnosis of hereditary pancreatitis (PRSS1 gene mutation)
* History of recurrent acute pancreatitis (>1 documented episode of characteristic abdominal pain associated with diagnostic imaging and/or elevated serum amylase or lipase > 3 times upper limit of normal).
* Pancreatic calcifications on CT scan
* At least 2 of the following:
* Endoscopic Ultrasound (EUS) with = or > 4 criteria for chronic pancreatitis (hyperechoic foci, strands, or ducts, lobulation, irregular duct margin, visible side - branches, calcifications, cysts, ductal dilatation) (28)
* Ductal (changes in side branch morphology) or parenchymal (loss of T1 signal intensity) abnormalities on secretin enhanced Magnetic resonance cholangiopancreatography (MRCP)
* Abnormal endoscopic pancreatic secretory function tests (HCO3 <= 75mmol/L at 30 or 45 minutes or <= 80mmol/L at 1 hour
* Subjects are capable of informed consent

Exclusion Criteria:

* Pregnancy
* Lactation
* Active acute pancreatitis or an episode of acute pancreatitis within 2 months of presentation for evaluation
* Pancreatic cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in pain scores based on Izbicki self-assessment score | Measured at weeks 0,4,6 and 10
  Difference in pain scores based on Izbicki self-assessment will be evaluated to determine if pancrelipase improves pain symptoms in patients with chronic pancreatitis

SECONDARY OUTCOMES:
Quality of life | Pancreatic Quality of Life Instrument (PANQOLI) assessment at weeks 0, 4, 6 and 10
  Difference in quality of live evaluated on PANQOLI assessment
Change in Narcotic Use | 0, 4, 6 and 10 weeks of treatment
  Difference in narcotic and non-narcotic use at 0, 4, 6 and 10 weeks of treatment as measured by morphine equivalents

CONTACTS AND LOCATIONS:
Overall Officials: Timothy B Gardner, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Yes
Within the confines of funding sponsors, and department of gastroenterology at Dartmouth

REFERENCES:
- [Background] Drewes AM, Krarup AL, Detlefsen S, Malmstrom ML, Dimcevski G, Funch-Jensen P. Pain in chronic pancreatitis: the role of neuropathic pain mechanisms. Gut. 2008 Nov;57(11):1616-27. doi: 10.1136/gut.2007.146621. Epub 2008 Jun 19. PMID 18566105
- [Background] Puylaert M, Kapural L, Van Zundert J, Peek D, Lataster A, Mekhail N, van Kleef M, Keulemans YC. 26. Pain in chronic pancreatitis. Pain Pract. 2011 Sep-Oct;11(5):492-505. doi: 10.1111/j.1533-2500.2011.00474.x. Epub 2011 Jun 16. PMID 21676159
- [Background] Kozarek RA, Ball TJ, Patterson DJ, Brandabur JJ, Traverso LW, Raltz S. Endoscopic pancreatic duct sphincterotomy: indications, technique, and analysis of results. Gastrointest Endosc. 1994 Sep-Oct;40(5):592-8. doi: 10.1016/s0016-5107(94)70260-8. PMID 7988825
- [Background] Bloechle C, Izbicki JR, Knoefel WT, Kuechler T, Broelsch CE. Quality of life in chronic pancreatitis--results after duodenum-preserving resection of the head of the pancreas. Pancreas. 1995 Jul;11(1):77-85. doi: 10.1097/00006676-199507000-00008. PMID 7667246
- [Background] Bellin MD, Freeman ML, Schwarzenberg SJ, Dunn TB, Beilman GJ, Vickers SM, Chinnakotla S, Balamurugan AN, Hering BJ, Radosevich DM, Moran A, Sutherland DE. Quality of life improves for pediatric patients after total pancreatectomy and islet autotransplant for chronic pancreatitis. Clin Gastroenterol Hepatol. 2011 Sep;9(9):793-9. doi: 10.1016/j.cgh.2011.04.024. Epub 2011 May 5. PMID 21683160
- [Background] Radnay PA, Brodman E, Mankikar D, Duncalf D. The effect of equi-analgesic doses of fentanyl, morphine, meperidine and pentazocine on common bile duct pressure. Anaesthesist. 1980 Jan;29(1):26-9. No abstract available. PMID 6104938
- [Background] Wilder-Smith CH, Hill L, Osler W, O'Keefe S. Effect of tramadol and morphine on pain and gastrointestinal motor function in patients with chronic pancreatitis. Dig Dis Sci. 1999 Jun;44(6):1107-16. doi: 10.1023/a:1026607703352. PMID 10389680
- [Background] Green GM, Lyman RL. Feedback regulation of pancreatic enzyme secretion as a mechanism for trypsin inhibitor-induced hypersecretion in rats. Proc Soc Exp Biol Med. 1972 May;140(1):6-12. doi: 10.3181/00379727-140-36384. No abstract available. PMID 5033119
- [Background] Ihse I, Lilja P, Lundquist I. Feedback regulation of pancreatic enzyme secretion by intestinal trypsin in man. Digestion. 1977;15(4):303-8. doi: 10.1159/000198016. PMID 863133
- [Background] Owyang C, Louie DS, Tatum D. Feedback regulation of pancreatic enzyme secretion. Suppression of cholecystokinin release by trypsin. J Clin Invest. 1986 Jun;77(6):2042-7. doi: 10.1172/JCI112534. PMID 3711342
- [Background] Slaff JI, Wolfe MM, Toskes PP. Elevated fasting cholecystokinin levels in pancreatic exocrine impairment: evidence to support feedback regulation. J Lab Clin Med. 1985 Mar;105(3):282-5. PMID 3973464
- [Background] Brown A, Hughes M, Tenner S, Banks PA. Does pancreatic enzyme supplementation reduce pain in patients with chronic pancreatitis: a meta-analysis. Am J Gastroenterol. 1997 Nov;92(11):2032-5. PMID 9362186
- [Background] Pancreatic Enzyme Supplementation for Treatment of Pain in Adult Patients with Chronic Pancreatitis: a Meta-Analysis and Systematic Review [abstract]. Gardner TB, Michalak D, Harrington MW, et al
- [Background] Slaff J, Jacobson D, Tillman CR, Curington C, Toskes P. Protease-specific suppression of pancreatic exocrine secretion. Gastroenterology. 1984 Jul;87(1):44-52. PMID 6202586
- [Background] Isaksson G, Ihse I. Pain reduction by an oral pancreatic enzyme preparation in chronic pancreatitis. Dig Dis Sci. 1983 Feb;28(2):97-102. doi: 10.1007/BF01315137. PMID 6825540
- [Background] Catalano MF, Sahai A, Levy M, Romagnuolo J, Wiersema M, Brugge W, Freeman M, Yamao K, Canto M, Hernandez LV. EUS-based criteria for the diagnosis of chronic pancreatitis: the Rosemont classification. Gastrointest Endosc. 2009 Jun;69(7):1251-61. doi: 10.1016/j.gie.2008.07.043. Epub 2009 Feb 24. PMID 19243769
- [Background] Zubarik R, Ganguly E. The rosemont criteria can predict the pain response to pancreatic enzyme supplementation in patients with suspected chronic pancreatitis undergoing endoscopic ultrasoun. Gut Liver. 2011 Dec;5(4):521-6. doi: 10.5009/gnl.2011.5.4.521. Epub 2011 Nov 21. PMID 22195253
- [Background] US Food and Drug Administration. FDA Approves Pancreatic Enzyme Replacement Product for Marketing in United States. Creon designed to help those with cystic fibrosis, others with exocrine pancreatic insufficiency. May 7th, 2009. Available at: http://www.fda.gov/NewsEvents/Newsroom/PressAnnouncements/ucm149579.htm
- [Background] Miyasaka K, Green GM. Effect of partial exclusion of pancreatic juice on rat basal pancreatic secretion. Gastroenterology. 1984 Jan;86(1):114-9. PMID 6689654
- [Background] Louie DS, May D, Miller P, Owyang C. Cholecystokinin mediates feedback regulation of pancreatic enzyme secretion in rats. Am J Physiol. 1986 Feb;250(2 Pt 1):G252-9. doi: 10.1152/ajpgi.1986.250.2.G252. PMID 3953805
- [Background] Lilja P. Effects of intraduodenal amylase, lipase, trypsin, and bile on pancreatic enzyme secretion in the rat. Eur Surg Res. 1980;12(6):383-91. doi: 10.1159/000128145. PMID 6167444
- [Background] Mossner J, Secknus R, Meyer J, Niederau C, Adler G. Treatment of pain with pancreatic extracts in chronic pancreatitis: results of a prospective placebo-controlled multicenter trial. Digestion. 1992;53(1-2):54-66. doi: 10.1159/000200971. PMID 1289173
- [Background] Winstead NS, Wilcox CM. Clinical trials of pancreatic enzyme replacement for painful chronic pancreatitis--a review. Pancreatology. 2009;9(4):344-50. doi: 10.1159/000212086. Epub 2009 May 18. PMID 19451744
- [Background] Waljee AK, Dimagno MJ, Wu BU, Schoenfeld PS, Conwell DL. Systematic review: pancreatic enzyme treatment of malabsorption associated with chronic pancreatitis. Aliment Pharmacol Ther. 2009 Feb 1;29(3):235-46. doi: 10.1111/j.1365-2036.2008.03885.x. Epub 2008 Nov 8. PMID 19035969
- [Background] Gullo L, Barbara L, Labo G. Effect of cessation of alcohol use on the course of pancreatic dysfunction in alcoholic pancreatitis. Gastroenterology. 1988 Oct;95(4):1063-8. doi: 10.1016/0016-5085(88)90184-9. PMID 3410221
- [Background] Midanik L. The validity of self-reported alcohol consumption and alcohol problems: a literature review. Br J Addict. 1982 Dec;77(4):357-82. doi: 10.1111/j.1360-0443.1982.tb02469.x. No abstract available. PMID 6762224
- [Background] Blondet JJ, Carlson AM, Kobayashi T, Jie T, Bellin M, Hering BJ, Freeman ML, Beilman GJ, Sutherland DE. The role of total pancreatectomy and islet autotransplantation for chronic pancreatitis. Surg Clin North Am. 2007 Dec;87(6):1477-501, x. doi: 10.1016/j.suc.2007.08.014. PMID 18053843
- [Background] Sahai AV, Zimmerman M, Aabakken L, Tarnasky PR, Cunningham JT, van Velse A, Hawes RH, Hoffman BJ. Prospective assessment of the ability of endoscopic ultrasound to diagnose, exclude, or establish the severity of chronic pancreatitis found by endoscopic retrograde cholangiopancreatography. Gastrointest Endosc. 1998 Jul;48(1):18-25. doi: 10.1016/s0016-5107(98)70123-3. PMID 9684659